CLINICAL TRIAL: NCT01586273
Title: Magnetic Resonance-guided High Intensity Focused Ultrasound for Palliation of Painful Skeletal Metastases - a Multicenter Study
Brief Title: Multicenter Study of Magnetic Resonance-guided High Intensity Focused Ultrasound for Pain Palliation of Bone Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 906273
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Bone Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MR-HIFU treatment (Experimental): Subjects undergo a MR-HIFU treatment for pain palliation of bone metastases on their most painful metastasis.
  Interventions: Device: MR-HIFU treatment for pain palliation of bone metastases

INTERVENTIONS:
Device: MR-HIFU treatment for pain palliation of bone metastases — A treatment session with the Philips Sonalleve MR-HIFU device for bone pain palliation with high-intensity focused ultrasound.
  Other Names: Philips Sonalleve MR-HIFU Bone Pain Palliative Therapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Philips Sonalleve Magnetic Resonance Imaging-guided High Intensity Focused Ultrasound (MR-HIFU) device for treating painful bone metastases.

DETAILED DESCRIPTION:
Magnetic Resonance Imaging-guided High Intensity Focused Ultrasound (MR-HIFU) is a non-invasive outpatient modality. In MR-HIFU, a specially designed ultrasound transducer is used to focus a beam of ultrasound energy into a small volume at a specific target site in the body. The focused beam is intended to produce therapeutic hyperthermia in the target field while only harmlessly warming the immediately surrounding tissue. Magnetic Resonance Imaging is used during the ultrasound treatment, both to focus the ultrasound beam on the target field and to perform real-time thermal mapping at and around the target.

The Philips Sonalleve MR-HIFU system is expected to be efficacious in reducing pain scores in patients with painful bone metastases and in reducing their pain medication usage.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with age ≥ 18 years
* Patient capable of giving informed consent and able to attend study visits
* Weight < 140kg
* Radiologic evidence of bone metastases from any solid tumor
* Diagnosis of dominant painful bone metastasis (Numerical Representative Scale (NRS) pain score ≥4), either refractory to standard of care (including radiotherapy and optimal pain medication) or standard of care is contra-indicated or refused by patient.
* Patient has been on stable pain medication for at least 1 week prior to HIFU treatment date
* Pain is localized to the targeted area, or is likely to be referred pain arising from the targeted area
* Patient has 1-3 painful lesions, and only the most painful lesion will be treated
* Intended Target Volume accessible for MR-HIFU procedure
* Target lesion maximum dimension ≤ 8cm
* Intended target volume visible by non-contrast MRI
* Distance between target and skin ≥ 1cm
* Patient is able to communicate sensation during MR-HIFU treatment
* MR-HIFU treatment date ≥ 4 weeks from last local treatment of the target lesion

Exclusion Criteria:

* Planned treatment lesion is a primary bone tumor or due to lymphoma, multiple myeloma, or leukemia.
* Communication barrier present
* Patient enrolled in another clinical study related to bone metastases treatment or pain relief treatment
* Unable to tolerate required stationary position during treatment
* Need for surgical stabilization in case of (impending) fracture (lytic lesion in weight-bearing bone larger than 50% of bone diameter)
* Pregnant woman
* Pain related to target lesion is predominantly due to fracture or impending fracture
* Pain related to target lesion is due to involvement of a neighboring major nerve by the metastatic tumor (cord or nerve compression)
* Target < 3cm from bladder / bowel / nerve along the beam path and < 1cm in the plane orthogonal to the beam
* Target in contact with hollow viscera
* Target located in skull, joints, ribs (when HIFU beam overlapping with lung), spine (excluding sacrum which is allowed) or sternum
* Scar along proposed HIFU beam path
* Internal or external fixation device along the proposed HIFU beam path or at the target
* MRI contraindicated (e.g. paramagnetic implants, pacemaker, claustrophobia)
* MRI contrast agent contraindicated (e.g. previous anaphylaxis or Glomerular Filtration Rate (GFR) < 30 ml/min/1.73m2)
* Sedation contraindicated
* Previous surgery or minimally invasive treatment at targeted site
* Clinically relevant medical history or abnormal physical findings that could interfere with the safety of the participant as judged by the treating physician or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pain response to therapy | 30 days after treatment
  Pain is measured using the Brief Pain Inventory (BPI) questionnaire. Patients are categorized into:
  * Complete response (CR): Pain score 0 without analgesic increase
  * Partial response (PR): Pain reduction of 2 or more without analgesic increase; or analgesic reduction of 25% without pain increase
  * Pain Progression (PP): Pain increase of 2 or more with stable analgesic use; or increase of 25% or more in analgesic use, with pain score stable or 1 point above baseline
  * No response corresponds to all other cases
  Patients with PR or CR at 30 days are considered responders to therapy.

SECONDARY OUTCOMES:
Total number of Adverse Events | within the first 90 days within treatment
  Total number of complications and adverse events, including the number of unintended lesions that occur as a result of treatment with MR-HIFU.
Quality of Life (as measured by questionnaire) | at day 0 before treatment, and at 7, 14, 30, 60 and 90 days after treatment
  Quality of Life will be measured at the given time points using a dedicated questionnaire for patients in palliative care: the European Organisation on Research and Treatment of Cancer (EORTC) C15-PAL questionnaire.
Subgroup analysis: pain response in radiation naïve patients | 30 days after treatment
  Assessment of positive response on pain (as determined by the Primary Outcome Measure) will be documented separately for radiation naïve patients and radiation failure patients, and a comparison between the two sub-groups will be performed.
Temporal evolution of pain response during the first 30 days after treatment | during the first 30 days after treatment
  Patients are given a diary to complete during the first 30 days after treatment, which documents their daily pain level on a 0-10 scale and their pain medication usage.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice A van den Bosch, MD, PhD, Principal Investigator — UMC Utrecht
Locations (3):
- University Medical Center Utrecht, Utrecht, Netherlands
- Samsung Medical Center, Seoul, South Korea
- Royal Marsden Hospital / Institute of Cancer Research, Sutton, Surrey, United Kingdom

REFERENCES:
- [Background] Catane R, Beck A, Inbar Y, Rabin T, Shabshin N, Hengst S, Pfeffer RM, Hanannel A, Dogadkin O, Liberman B, Kopelman D. MR-guided focused ultrasound surgery (MRgFUS) for the palliation of pain in patients with bone metastases--preliminary clinical experience. Ann Oncol. 2007 Jan;18(1):163-167. doi: 10.1093/annonc/mdl335. Epub 2006 Oct 9. PMID 17030549
- [Background] Gianfelice D, Gupta C, Kucharczyk W, Bret P, Havill D, Clemons M. Palliative treatment of painful bone metastases with MR imaging--guided focused ultrasound. Radiology. 2008 Oct;249(1):355-63. doi: 10.1148/radiol.2491071523. Epub 2008 Aug 11. PMID 18695209
- [Background] Liberman B, Gianfelice D, Inbar Y, Beck A, Rabin T, Shabshin N, Chander G, Hengst S, Pfeffer R, Chechick A, Hanannel A, Dogadkin O, Catane R. Pain palliation in patients with bone metastases using MR-guided focused ultrasound surgery: a multicenter study. Ann Surg Oncol. 2009 Jan;16(1):140-6. doi: 10.1245/s10434-008-0011-2. Epub 2008 Nov 11. PMID 19002530
- [Background] Chow E, Hoskin P, Mitera G, Zeng L, Lutz S, Roos D, Hahn C, van der Linden Y, Hartsell W, Kumar E; International Bone Metastases Consensus Working Party. Update of the international consensus on palliative radiotherapy endpoints for future clinical trials in bone metastases. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1730-7. doi: 10.1016/j.ijrobp.2011.02.008. Epub 2011 Apr 12. PMID 21489705
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Groenvold M, Petersen MA, Aaronson NK, Arraras JI, Blazeby JM, Bottomley A, Fayers PM, de Graeff A, Hammerlid E, Kaasa S, Sprangers MA, Bjorner JB; EORTC Quality of Life Group. The development of the EORTC QLQ-C15-PAL: a shortened questionnaire for cancer patients in palliative care. Eur J Cancer. 2006 Jan;42(1):55-64. doi: 10.1016/j.ejca.2005.06.022. Epub 2005 Sep 12. PMID 16162404
- [Background] Chow E, Hird A, Velikova G, Johnson C, Dewolf L, Bezjak A, Wu J, Shafiq J, Sezer O, Kardamakis D, van der Linden Y, Ma B, Castro M, Arnalot PF, Ahmedzai S, Clemons M, Hoskin P, Yee A, Brundage M, Bottomley A; EORTC Quality of Life Group. The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for patients with bone metastases: the EORTC QLQ-BM22. Eur J Cancer. 2009 May;45(7):1146-1152. doi: 10.1016/j.ejca.2008.11.013. Epub 2008 Dec 25. PMID 19097882